CLINICAL TRIAL: NCT02597608
Title: Impact Evaluation of the DFID Programme to Accelerate Improved Nutrition of the Extreme Poor in Bangladesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Food Policy Research Institute (Other)
Collaborators: Department for International Development, United Kingdom (Other Government); Institute of Development Studies (Other); Chars Livelihoods Programme (Other); Shiree, Stimulating Household Improvements Resulting in Economic Empowerment (Other); Urban Partnerships for Poverty Reduction (Other); Consortium of International Agricultural Research Centers (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 601059.001.001
Record Dates: First submitted 2015-10-28; First posted 2015-11-05 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2015-11

CONDITIONS: Child Nutritional Status; Household Dietary Diversity; Maternal Nutrition Knowledge and Practices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- UPPR: Control (Experimental): No interventions are provided.
  Interventions: Other: UPPR: Control
- UPPR: Livelihoods only (Experimental): Livelihoods programmes offered by UPPR.
  Interventions: Behavioral: UPPR: Livelihoods
- UPPR: Livelihoods plus nutrition (Experimental): Livelihoods programmes offered by UPPR, plus nutrition programmes offered by UPPR.
  Interventions: Behavioral: UPPR: Livelihoods; Dietary Supplement: UPPR: Nutrition
- CLP: Livelihoods only (Experimental): Livelihoods programmes offered by CLP.
  Interventions: Behavioral: CLP: Livelihoods
- CLP: Livelihoods plus nutrition (Experimental): Livelihoods programmes offered by CLP, plus nutrition programmes offered by CLP.
  Interventions: Behavioral: CLP: Livelihoods; Dietary Supplement: CLP: Nutrition
- Shiree: Livelihoods only (Experimental): Livelihoods programmes offered by Shiree.
  Interventions: Behavioral: Shiree: Livelihoods
- Shiree: Livelihoods plus nutrition (Experimental): Livelihoods programmes offered by Shiree, plus nutrition programmes offered by Shiree.
  Interventions: Behavioral: Shiree: Livelihoods; Dietary Supplement: Shiree: Nutrition

INTERVENTIONS:
Behavioral: CLP: Livelihoods — Capital for purchase of income generating asset, physical infrastructure (plinths, latrines, tubewells), livelihood maintenance stipend, monthly asset maintenance cost stipend, agricultural livelihood training, non-agricultural livelihood training, financial training, health and nutrition training.
  Arms: CLP: Livelihoods only; CLP: Livelihoods plus nutrition
Dietary Supplement: CLP: Nutrition — Counseling on breastfeeding and complementary feeding; five components micronutrients (iron 12.5 mg, folic acid 0.16 mg, zinc 5 mg, vitamin A 0.3 mg, vitamin C 30 mg) for children 7-23 months dosage of 120 sachets per year; 180 iron and folic acid tablets (60 mg iron and 400 mg folic acid) tablets to each pregnant woman after first trimester and up to 180 for each breastfeeding woman per year, as well as 104 tablets to each adolescent girl; deworming treatment for children aged 1-5 years, adolescent girls, pregnant women after first trimester; identification and referral of acute malnutrition; facilitation of government campaigns on nutrition.
  Arms: CLP: Livelihoods plus nutrition
Behavioral: Shiree: Livelihoods — Financial training; input support for livelihoods (cropping, livestock, poultry, fishing, bamboo working, small businesses, tailoring etc.); capacity building (mobilising Self Help Groups, facilitating community based organizations (CBOs), skills transfer); innovation support (market linkage and access to value chains); credit and savings groups; support in mobilizing communities to advocate for their needs.
  Arms: Shiree: Livelihoods only; Shiree: Livelihoods plus nutrition
Dietary Supplement: Shiree: Nutrition — Counseling on breastfeeding, complementary feeding, and sanitation; community discussions including adolescent girls on early and forced marriage; five components micronutrients (iron 12.5 mg, folic acid 0.16 mg, zinc 5 mg, vitamin A 0.3 mg, vitamin C 30 mg) for children aged 7-23 months; 180 iron and folic acid tablets (60 mg iron and 400 mg folic acid) tablets to each pregnant woman after first trimester and up to 180 for each breastfeeding woman per year, as well as 104 tablets to each adolescent girl; deworming treatment for children aged 1-5 years, adolescent girls, pregnant women after first trimester.
  Arms: Shiree: Livelihoods plus nutrition
Behavioral: UPPR: Livelihoods — Monetary support for communities to improve infrastructure (drains, footpaths, latrines and water dwells, access to roads and markets); financing for apprenticeships; grants for small businesses; education grants for girls; grants for urban food production activities; financial training; establishment of savings and credit groups; support for communities in advocating for their needs; microcredit; improving access to health facilities; improving housing conditions; provision of plinths.
  Arms: UPPR: Livelihoods only; UPPR: Livelihoods plus nutrition
Dietary Supplement: UPPR: Nutrition — Counseling on breastfeeding, complementary feeding, and sanitation; community discussions including adolescent girls on early and forced marriage; five components micronutrients (iron 12.5 mg, folic acid 0.16 mg, zinc 5 mg, vitamin A 0.3 mg, vitamin C 30 mg) for children aged 7-23 months; 180 iron and folic acid tablets (60 mg iron and 400 mg folic acid) tablets to each pregnant woman after first trimester and up to 180 for each breastfeeding woman per year, as well as 104 tablets to each adolescent girl; deworming treatment for children aged 1-5 years, adolescent girls, pregnant women after first trimester.
  Arms: UPPR: Livelihoods plus nutrition
Other: UPPR: Control — No interventions provided.
  Arms: UPPR: Control

SUMMARY:
This is a randomized study in three areas of Bangladesh (Chars region where CLP operates, Haor region where Shiree operates, and urban slums where UPPR operates). Treatment is assigned at the community level, where treatments are:

* Livelihoods intervention only (L only)
* Livelihoods intervention plus nutrition intervention (L+N)

In UPPR only, the study also includes a non-randomly selected comparison group (C).

Within treatment localities, targeted beneficiaries include women, adolescent girls, and children under 24 months. Benefits are received for two years.

DETAILED DESCRIPTION:
Undernutrition is widespread in Bangladesh. In 2011, according to the Bangladesh Demographic and Health Survey, 41.3 per cent of children under age five were stunted, 36.4 per cent were underweight, 15.6 per cent were wasted, and more than 50 per cent were anaemic. Prevalences were even higher among extremely poor households. Meanwhile, evidence from South Asia shows that high rates of economic growth and reduction in poverty have not led to similarly large reductions in undernutrition (see 1, 2, 3). These findings have suggested that improvements in income alone may not be sufficient to improve nutritional status. Extensive research has also shown that the critical window for nutritional interventions is during the "first thousand days" of life (see 4, 5), from the time when a child is in utero until about two years of age. Based on this accumulated evidence, growing attention has come to introducing nutrition interventions that target children's "first thousand days" alongside household poverty reduction programmes. In particular, there has been growing emphasis on nutrition interventions that aim to improve infant and young child feeding practices-through increasing nutritional knowledge of women who are pregnant, lactating, or likely to be pregnant in the future-as well as to improve the nutritional status of these women themselves.

Although there exists considerable evidence assessing the effectiveness of various livelihoods interventions and other social protection programmes, as well as some evidence on the effectiveness of various direct nutritional interventions, little research directly assesses how an integrated livelihoods and nutrition programme might compare with livelihoods support alone. There are several reasons why the combination of nutrition and livelihoods support may have nutritional benefits over and above livelihoods support only. First, a key constraint to improved nutritional status may be insufficient knowledge of appropriate infant and young child feeding practices (for example, the appropriate duration of exclusive breastfeeding, the appropriate frequency and diversity of child feeding thereafter, etc.). If this is the case, then improving income alone will not necessarily lead to improved feeding practices. Second, there may be synergies between the two types of support. For example, even if a mother's knowledge of infant and young child feeding practices improves, she may still need access to sufficient resources for undertaking those practices (such as income to purchase the recommended types of food), which can be facilitated through a livelihoods intervention. Third, there may be other dynamics shifted through the direct nutrition intervention that mediate how the livelihoods intervention affects nutritional status. For example, if a direct nutrition intervention targeting women improves women's bargaining power within the household, and if women tend to prefer devoting more resources to young children's nutrition (e.g., Quisumbing and Maluccio 2003), the result may also be larger impacts on nutritional status than livelihoods support alone.

The DFID Programme to Accelerate Improved Nutrition for the Extreme Poor in Bangladesh aims to improve nutrition outcomes for young children, pregnant and lactating mothers, and adolescent girls. Its approach is to integrate direct nutrition interventions into the livelihood support currently provided to extremely poor households in Bangladesh through three existing programmes: the Chars Livelihoods Programme (CLP), the Shiree Economic Empowerment of the Poorest Programme (Shiree or EEP, within which the investigators focus on the Concern subproject), and the Urban Partnership for Poverty Reduction Programme (UPPR).

In order to rigorously and independently assess the impacts of these integrated nutrition and livelihoods programmes, DFID has collaborated with research partners and implementation partners to undertake a mixed methods impact evaluation, entitled "Impact Evaluation of the DFID Programme to Accelerate Improved Nutrition for the Extreme Poor in Bangladesh." The evaluation team includes IDS (the lead organisation), IFPRI, ITAD, CNRS, and BRAC University. The evaluation uses mixed quantitative and qualitative methods within a strong theory-based design to assess the impacts of the integrated programmes on nutritional status.

The quantitative impact component involves a baseline survey (conducted in September-November 2013) and an endline survey (to be conducted in November-December 2015). The exploratory/explanatory component includes a qualitative subcomponent (for which the first phase of fieldwork has been ongoing since February 2014), as well as a process evaluation subcomponent (ongoing since July 2014, final results not yet available). The cost effectiveness component began in August 2014 and will be completed in early 2016 following the quantitative endline survey completion.

The three key research questions regarding programme impact that will be addressed are:

1. What is the impact on nutrition outcomes of receiving a combination of livelihoods and direct nutrition interventions (denoting this scenario (L+N)), relative to receiving a livelihoods intervention only (denoting this scenario (L))?
2. What is the impact on nutrition outcomes of receiving a combination of livelihoods and direct nutrition interventions (L+N), relative to receiving no intervention (denoting this scenario (C) for control)?
3. What is the impact on nutrition outcomes of receiving a livelihoods intervention only (L), relative to receiving no intervention (C)? This will pertain only to the urban group served by UPPR.

In order to construct a proxy for the (L+N) households in the counterfactual (L) scenario, randomisation is used. Among the households that already receive the livelihoods intervention at baseline, half are randomly assigned to additionally receive the nutrition intervention after the baseline (denoted the (L+N) group). The remaining half continue to receive only the livelihoods intervention (denoting the (L) group). Randomisation is conducted at the level of primary sampling units (PSUs) that cover an entire locality, rather than at the level of individual households. The randomisation makes it very likely that characteristics of the (L) and (L+N) groups will on average be similar at baseline. (L) is then a valid proxy for (L+N), and average differences between the groups at endline can be interpreted as impacts caused only by the addition of the nutrition component rather than pre-existing differences.

In order to construct a proxy for the (L+N) households in the counterfactual (C) scenario of no intervention, non-randomised approaches are used. Since none of the original livelihoods interventions was rolled out following a randomised control trial design, there is no obvious set of comparable non-beneficiaries to serve as the counterfactual. Because a control group is nonetheless required to assess the absolute benefits of either (L) or (L + N) interventions, attempts were made to construct the best possible control group out of non-randomly selected non-beneficiaries. It is important to emphasise that a non-random control group is not expected to be on average identical to beneficiary households. In the baseline survey, the objective was simply to sample a group of non-beneficiaries as similar as possible to the beneficiaries except for receipt of the intervention.

Major topics areas covered by the qualitative data collection tools include the following:

1. Social, economic, institutional and political context of the community
2. Local practices, resources, customs in regards to health, hygiene, nutrition and care of children, pregnant and lactation mothers, adolescent girls
3. For (L) and (L+N) sites: Perceived impact of the livelihood intervention
4. For (L+N) sites: Perceived synergies and disconnects between the nutrition and livelihood interventions in the communities
5. For (L+N) sites: Micro-dynamics of the nutrition intervention at the community level and how beneficiaries perceive/experience the intervention

ELIGIBILITY:
Inclusion Criteria:

* Children (boys and girls) 0-36 months
* Pregnant and breastfeeding women
* Adolescent girls (aged 13-19)
* Households must meet eligibility criteria of each of the three programmes (CLP, Shiree, UPPR) except for the control group in UPPR.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 11340 (Actual)
Dates: Start 2013-07; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Child anthropometry - height for age | Baseline. Up to 24 months.
  Height for age z scores. Outcomes specified in terms of levels two years after intervention started, as well as in changes (2013-2015).
Child food intake - number unique foods | Baseline. Up to 24 months.
  Number of unique foods consumed in previous 24 hours. Outcomes specified in terms of levels two years after intervention started, and as changes (2013-2015).
Dietary diversity of index child's mother, father, and of adolescent girl - unique foods | Baseline. Up to 24 months.
  Number of unique foods consumed in previous 24 hours. Outcomes specified in terms of levels two years after intervention started, and as changes (2013-2015).
Index child mother's nutrition knowledge | Baseline. Up to 24 months.
  Knowledge (total score) of index child's mother regarding questions on breastfeeding, complementary feeding, nutrition, and sanitation practices (29 questions). Outcomes specified in terms of levels two years after intervention started, and as changes (2013-2015).
Household food security - food groups | Baseline. Up to 24 months.
  Food groups consumed by household in previous seven days. Outcomes specified in terms of levels two years after intervention started, and as changes (2013-2015).
Infant and young child feeding practices - breastfeeding | Baseline. Up to 24 months.
  Length of breastfeeding of index child. Outcomes specified in terms of levels two years after intervention started, and as changes (2013-2015).
Receipt of and participation in livelihoods and nutrition interventions (take up) | Baseline. Up to 24 months.
  Whether received livelihoods and nutrition interventions carried out by CLP/Shiree/UPPR programmes. Outcomes specified in terms of levels two years after intervention started, and as changes (2013-2015).
Community nutrition worker knowledge and activities. | Up to 24 months.
  Misconceptions regarding nutrition knowledge and attitudes (regarding breastfeeding, complementary feeding, and sanitation knowledge). Outcomes specified in terms of levels two years after intervention started.
Child anthropometry - weight for age | Baseline. Up to 24 months.
  Weight for age z scores. Outcomes specified in terms of levels two years after intervention started, as well as in changes (2013-2015).
Child anthropometry - stunting | Baseline. Up to 24 months.
  Percentage of children 0-24 stunted. Outcomes specified in terms of levels two years after intervention started, as well as in changes (2013-2015).
Child anthropometry - wasting | Baseline. Up to 24 months.
  Percentage of children 0-24 wasted. Outcomes specified in terms of levels two years after intervention started, as well as in changes (2013-2015).
Child food intake - number food groups | Baseline. Up to 24 months.
  Number of food groups consumed in previous 24 hours. Outcomes specified in terms of levels two years after intervention started, and as changes (2013-2015).
Child food intake - food groups | Baseline. Up to 24 months
  Consumption of specific food groups (animal source foods, dairy, vitamin A rich foods, etc.) in previous 24 hours. Outcomes specified in terms of levels two years after intervention started, and as changes (2013-2015).
Child food intake - caloric consumption | Baseline. Up to 24 months.
  Caloric consumption in previous 24 hours. Outcomes specified in terms of levels two years after intervention started, and as changes (2013-2015).
Dietary diversity of index child's mother, father, and of adolescent girl | Baseline. Up to 24 months.
  Number of food groups consumed in previous 24 hours. Outcomes specified in terms of levels two years after intervention started, and as changes (2013-2015).
Household food security - unique foods | Baseline. Up to 24 months.
  Number of unique foods consumed in previous seven days. Outcomes specified in terms of levels two years after intervention started, and as changes (2013-2015).
Household food security - number of food groups | Baseline. Up to 24 months.
  Number of food groups consumed in previous seven days weighted by nutritional value and frequency of consumption. Outcomes specified in terms of levels two years after intervention started, and as changes (2013-2015).
Household food security - value of consumption | Baseline. Up to 24 months.
  Value of food consumption in previous seven days. Outcomes specified in terms of levels two years after intervention started, and as changes (2013-2015).
Household food security - caloric availability | Baseline. Up to 24 months.
  Household caloric availability in previous seven days. Outcomes specified in terms of levels two years after intervention started, and as changes (2013-2015).
Infant and young child feeding practices - complementary feeding | Baseline. Up to 24 months.
  Age complementary feeding initiated. Outcomes specified in terms of levels two years after intervention started, and as changes (2013-2015).
Community nutrition worker knowledge and activities | Up to 24 months.
  Number of home visits and group training sessions in past month. Outcomes specified in terms of levels two years after intervention started.
Child anthropometry - weight for height | Baseline. Up to 24 months.
  Weight for height z scores. Outcomes specified in terms of levels two years after intervention started, as well as in changes (2013-2015).
Women's BMI | Baseline. Up to 24 months.
  Body mass index of index child's mother. Weight for height z scores. Outcomes specified in terms of levels two years after intervention started, as well as in changes (2013-2015).

SECONDARY OUTCOMES:
Nutrition knowledge of adolescent girl | Baseline. Up to 24 months.
  Knowledge (total score out of 29) of adolescent girl regarding breastfeeding, complementary feeding, nutrition, and sanitation practices (29 questions). Outcomes specified in terms of levels two years after intervention started, and as changes (2013-2015).
Health of index child <36 months - child ill | Baseline. Up to 24 months.
  Did mother report child was ill in previous 2 weeks. Outcomes specified in terms of levels two years after intervention started, and as changes (2013-2015).
Antenatal care - attendance | Baseline. Up to 24 months.
  Attendance at antenatal care sessions. Outcomes specified in terms of levels two years after intervention started, and as changes (2013-2015).
Sanitation practices for index child | Baseline. Up to 24 months.
  Disposal of stool of index child. Outcomes specified in terms of levels two years after intervention started, and as changes (2013-2015).
Women's status index | Baseline. Up to 24 months.
  Index constructed using principal components analysis (including: ability to work, decision making power in spending earnings, decision making power in household expenditures, mobility outside the household, participation in group meetings, voting, respect and domestic violence, control and agency, time preferences). Outcomes specified in terms of levels two years after intervention started, and as changes (2013-2015).
Ownership of assets - value | Baseline. Up to 24 months.
  Value of total assets owned. Outcomes specified in terms of levels two years after intervention started, and as changes (2013-2015).
Housing quality | Baseline. Up to 24 months.
  Index using principal components analysis including: ownership status of house, quality of materials of house, electricity and fuel sources, acquisition of plinths, water and sanitation quality. Outcomes specified in terms of levels two years after intervention started, and as changes (2013-2015).
Household consumption - food consumption | Baseline. Up to 24 months.
  Value of food consumption in previous seven days. Outcomes specified in terms of levels two years after intervention started, and as changes (2013-2015).
Household income | Baseline. Up to 24 months.
  Value of annual total income derived from all sources. Outcomes specified in terms of levels two years after intervention started, and as changes (2013-2015).
Health of index child <36 months - care sought | Baseline. Up to 24 months.
  Whether care was sought. Outcomes specified in terms of levels two years after intervention started, and as changes (2013-2015).
Health of index child < 36 months - where care received | Baseline. Up to 24 months.
  Where care was received. Outcomes specified in terms of levels two years after intervention started, and as changes (2013-2015).
Antenatal care | Baseline. Up to 24 months.
  Care received at antenatal sessions (total score on receipt of food, and receipt of iron folic acid and vitamin A tablets). Outcomes specified in terms of levels two years after intervention started, and as changes (2013-2015).
Care at birth | Baseline. Up to 24 months.
  Care received at antenatal sessions (total score on location of delivery of index child, weighing of index child after birth). Outcomes specified in terms of levels two years after intervention started, and as changes (2013-2015).
Household consumption - value of non-food consumption | Baseline. Up to 24 months.
  Value of monthly non-food consumption. Outcomes specified in terms of levels two years after intervention started, and as changes (2013-2015).
Household consumption - value of non-food consumption subgroups | Baseline. Up to 24 months.
  Value of monthly non-food consumption by specified sub-groups (clothing, medical expenses, education expenses, transport, consumables, semi-durables). Outcomes specified in terms of levels two years after intervention started, and as changes (2013-2015).
Household consumption - food and non-food | Baseline. Up to 24 months.
  Value of monthly total household consumption (food and non-food). Outcomes specified in terms of levels two years after intervention started, and as changes (2013-2015).

CONTACTS AND LOCATIONS:
Overall Officials: John Hoddinott, DPhil, Principal Investigator — Cornell University; Shalini Roy, PhD, Principal Investigator — International Food Policy Research Institute; Naureen Karachiwalla, DPhil, Principal Investigator — International Food Policy Research Institute; Firdousi Naher, PhD, Principal Investigator — University of Dhaka; Nick Nisbett, PhD, Principal Investigator — Institute for Development Studies, University of Sussex; Jean Pierre Tranchant, PhD, Principal Investigator — Institute for Development Studies, University of Sussex
Locations (1):
- International Food Policy Research Institute, Dhaka, Bangladesh

REFERENCES:
- [Background] Smith, L. C., U. Ramakrishnan, A. Ndiaye, L. Haddad, and R. Martorell. 2002. "The Asian Engima. Chapter 7 of The Importance of Women's Status for Child Nutrition in Developing Countries. Research Report 131. Washington, DC: International Food Policy Research Institute.
- [Background] Ramalingaswami, V., U. Jonsson, and J. Rohde. 1996. "Commentary: The Asian Enigma." In The Progress of Nations. New York: UNICEF.
- [Background] Deaton, A., and J. Dreze. 2009.
- [Background] Bhutta ZA, Das JK, Rizvi A, Gaffey MF, Walker N, Horton S, Webb P, Lartey A, Black RE; Lancet Nutrition Interventions Review Group, the Maternal and Child Nutrition Study Group. Evidence-based interventions for improvement of maternal and child nutrition: what can be done and at what cost? Lancet. 2013 Aug 3;382(9890):452-477. doi: 10.1016/S0140-6736(13)60996-4. Epub 2013 Jun 6. PMID 23746776
- [Background] Hoddinott J, Behrman JR, Maluccio JA, Melgar P, Quisumbing AR, Ramirez-Zea M, Stein AD, Yount KM, Martorell R. Adult consequences of growth failure in early childhood. Am J Clin Nutr. 2013 Nov;98(5):1170-8. doi: 10.3945/ajcn.113.064584. Epub 2013 Sep 4. PMID 24004889